CLINICAL TRIAL: NCT07007507
Title: Attendance and Adherence to Aerobic Exercise After Subacute Stroke: A Pilot Study
Brief Title: Attendance and Adherence to Aerobic Exercise After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ostergotland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Klas Sandberg, PhD. PT, Ostergotland County Council, Sweden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024-04914-01
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: Stroke, Aerobic exercise, Attendence, Adherence
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aerobic Exercise (Experimental): Two organized training sessions per week and one personal fitness activity once a week
  Interventions: Behavioral: Aerobic Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — Aerobic exercise is performed by repeating sequences of light to moderate intensity activities for extended periods of time.(12) The American Heart Association recommends that for stroke survivors, exercise intensity should be 40%-70% of VO2 reserve or heart rate (HR) reserve; 55%-80% HR max; RPE 11-14 Borg rating of perceived exertion (RPE) scale 6-20 scale, 3-5 days/week, 30-60 min/session (or multiple 10 min sessions)

SUMMARY:
Stroke is a common cause of functional impairment and a disease that requires large financial resources and days of care(1). For a few years now, group or individual cardiorespiratory training has been a recommended part of subacute rehabilitation after stroke(2). The training form should be a routine part of stroke rehabilitation and should be able to be carried out in both hospitals, municipal facilities and at home(2). The benefits include better walking ability and improved quality of life(3). Despite the possible benefits of cardiorespiratory training, access to the training form has been limited and compliance with the recommendations has been low(4). The Rehab East Neuro Unit has decided to implement the training form in the spring of 2024 to increase access to the training form after stroke.

The purpose of this pilot study is to study attendance at training sessions and adherence with the training form's recommendations and guidelines over a six-month period.

By identifying any challenges that may arise during the study with recruitment, retention of participants or data collection, the pilot study will form the basis for a larger study that will involve multiple study sites. The pilot study will, through study protocols and interviews or surveys of patients and staff, shed light on study design, instruments for data collection and analysis methods. The results will be used to ensure that further studies are effective, appropriate and feasible. Compliance with guidelines will be evaluated with an exercise diary or digital registration.

DETAILED DESCRIPTION:
Background During the last decades, various forms of exercise after stroke have been proposed(6). In 2000, cardiorespiratory exercise had a breakthrough when neurorehabilitation was introduced as a new field of research. Swedish research showed that neurons are capable of neurogenesis and plasticity(7,8). Experimental studies showed that exercise could be an important catalyst in this process.(9) Interest in fitness training after stroke was soon reflected in major reviews with a rapidly increasing number of published articles (10). Exercise is described as a range of physical activity that is planned, structured, and repetitive and has improvement or maintenance of physical fitness as an intermediate or ultimate goal.(11) Aerobic exercise refers to the use of oxygen in the combustion to adequately meet the energy demand during exercise via aerobic metabolism.(12) Aerobic exercise is performed by repeating sequences of activities with light to moderate intensity for extended periods of time.(12) The American Heart Association recommends for stroke survivors that exercise intensity should be 40%-70% of Vo2 reserve or heart rate (HR) reserve; 55%-80% HR max; RPE 11-14 Borg rating of perceived exertion (RPE) scale 6-20 scale, 3-5 days/week, 30-60 min/session (or several 10-minute sessions)(13) Studies have shown that cardiorespiratory exercise can affect recovery after stroke. The mechanisms behind the improvement have not been fully elucidated, but the form of exercise can be expected to affect healing after the injury. Cardiorespiratory exercise in groups or individually has been a recommended part of subacute rehabilitation after stroke for a few years(2). Despite the possible benefits of cardiorespiratory exercise, access to the form of exercise has been limited and compliance with the recommendations has been low(4). Identification of barriers to the form of exercise is of great importance in order to be able to offer optimal recovery opportunities for the disease group. There is currently a lack of studies on how many patients participate in the form of exercise or how many patients reach the recommendations.

Purpose - question Primary purpose: The purpose of the pilot study is to study and evaluate participation and adherence to group-based fitness training in the subacute phase after stroke. The work also aims to study and test methods for studying the patient's experiences with the training and factors that affect the implementation of the training in everyday clinical practice

The purpose of the pilot study is to study attendance at training sessions and adherence to the training format's recommendations and guidelines over a period of six months.

* To investigate how many patients are willing to participate in fitness-based group training after stroke.
* To investigate how many of these patients reach the recommended amount and intensity of training.
* To investigate the patient's experiences with the training format

Method The pilot study is conducted as a prospective cohort study at Vrinnevis Hospital's stroke unit. Patients are invited consecutively after becoming ill and completing inpatient care. The invitation to training is made by the responsible physiotherapist in consultation with the responsible physician. Training starts after discharge and no earlier than 7 days after illness and up to and including 6 months after illness. Training sessions and training program are designed so that current guidelines can be achieved. Two training sessions are offered at Vrinnvis Hospital under the guidance of a physiotherapist. Additional training sessions are carried out at home according to an individually designed program by a physiotherapist. Descriptive statistics are used to describe individual variables and attendance.

All stroke patients who are able to walk 5 meters and can sit on an ergometer cycle are invited. NIHSS 6

Patients with medical or orthopedic problems that prevent the implementation of training should not participate in the study.

Study participants must be able to read and understand the Swedish language in order to be able to assimilate study information

The study will be carried out close to the usual clinical routine after stroke and only a few outcome variables and study-specific forms will be added.Study start: September 2024 and the pilot study is expected to last until April 2025.

After the training period, training diaries and registered training sessions will be documented in a study-specific database and analyzed for attendance and compliance. To achieve 100% compliance with the guidelines, the patient must complete a total of 3 training sessions of 30-60 minutes per week for 12 weeks. Interviews or surveys of the patients' experience of the training will be conducted after the training has been completed after week 12.

ELIGIBILITY:
Inclusion Criteria:

All stroke patients who can walk 5 meters and can sit on an ergometer cycle are invited.- Study participants must be able to read and understand the Swedish language in order to be able to assimilate study information.

Exclusion Criteria:

Patients with medical or orthopedic conditions that prevent exercise should not participate in the study.-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Attendence | From enrollment to the end of treatment after 8 weeks
  Participation in number of organized training sessions and own physical activities

SECONDARY OUTCOMES:
Adherence | From enrollment to the end of treatment after 8 weeks
  To achieve 100% adherence with the guidelines, the patient must complete a total of 3 training sessions of 30-60 minutes per week for 8 weeks. Interviews or surveys of the patients' experience of the training will be conducted after the training has been completed after week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Klas Sandberg, PhD, Principal Investigator — Ostergotland CC; Klas Sandberg, PhD, Study Director — Ostergotland CC
Locations (1):
- Vrinnevisjukhuset, Norrköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
This is a pilotstudy with focus on feasability. Further, in a large full scale study maybe IPD will be shared.